CLINICAL TRIAL: NCT06315816
Title: The Effect of Virtual Reality Glasses Used During Tooth Extraction and Extirpation Treatment Under Local Anesthesia on Anxiety and Fear in 7-10 Years Old Children
Brief Title: Virtual Reality Used During Tooth Extraction and Extirpation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murat Bektaş (Other)
Responsible Party: Sponsor-Investigator, Murat Bektaş, Head of Department, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DokuzEU-1
Record Dates: First submitted 2023-12-29; First posted 2024-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Anxiety and Fear; Tooth Disease
Keywords: Tooth extraction; Extirpation; Child; Anxiety; fear; Nursing; virtual reality
MeSH Terms: conditions — Anxiety Disorders; Tooth Diseases

STUDY DESIGN:
Intervention Model Description: The population will consist of children between the ages of 7-10 who presented to the pediatric dental clinic of an oral and dental health center Turkey. The sample size of the study was calculated as GPOWER 3.1 statistical analysis software, based on a significance level of 0.05, a power value of 80%, and an effect size of 0.15 (medium effect size). Considering 10% attrition, it will plan to sample a total of 80 children, including 40 in the experimental group and 40 in the control group. Eventually, a total of 120 children, 60 in the experimental group and 60 in the control group,will include in the study to reveal the relationship between the variables more clearly.
Who Masked: Outcomes Assessor
Masking Description: The data will be analyzed by a statistician blind to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal (Experimental): The children will ask to choose a three-dimensional cartoon from the list to watch during the procedure, it will run, the mobile phone will placed into the virtual reality glasses, and the children wear the VR glasses and start watching the cartoon. During the procedure, the children's parents and the researcher will present, and the children watch the cartoon through virtual reality glasses. After the procedure, the virtual reality glasses will removed, and ten minutes after the procedure will completed, the CFS and the CAS-S will apply as a post-test.
  Interventions: Behavioral: virtual reality glasses used during tooth extraction and extirpation treatment
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: virtual reality glasses used during tooth extraction and extirpation treatment — The effect of virtual reality glasses used during tooth extraction and extirpation treatment under local anesthesia on anxiety and fear in 7-10 years old children
  Arms: Experimantal

SUMMARY:
This study carriy out to evaluate the effect of virtual reality glasses used during tooth extraction and extirpation treatment under local anesthesia on anxiety and fear in children aged 7-10 years.

DETAILED DESCRIPTION:
Aims and Objectives: Virtual reality glasses can be used as a distraction method in dental practices for children. This study carriy out to evaluate the effect of virtual reality glasses used during tooth extraction and extirpation treatment under local anesthesia on anxiety and fear in children aged 7-10 years.

Design: A randomized controlled experimental study design will use. Methods: The sample of the study consisted of 120 seven to ten-year-old children, including 60 in the experimental group and 60 in the control group, who will receive tooth extraction and extirpation treatment in the pediatric dental clinic of an oral and dental health center. Data collection tools included a Child and Family Information Form, the Children's Fear Scale, and the Child Anxiety Scale-State. During the procedure, the children in the experimental group will watch a video that they chose through virtual reality glasses. No intervention will apply to the control group. Data will analyz using the Chi-square test, t-test, Shapiro-Wilk, mean, and percentage distributions.

ELIGIBILITY:
Inclusion Criteria:

* Children who will between the ages of 7-10,
* Children who have Tooth Extraction
* Children who have Extirpation Treatment
* Have no cognitive development problems,

Exclusion Criteria:

* Children who will not want to participate in the study,
* Leave the research during the study,
* Have an audio-visual disorder that could prevent the use of virtual glasses.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety Means | 1-4 Weeks
  Anxiety score will be measured with the Child Fear and Anxiety Scale. The lowest score from the scale can be 0 and the highest score can be 10. As the score obtained from the scale increases, the child's anxiety increases. In this study, if children get high scores from the anxiety section of the scale, it will be determined that they have high procedural anxiety. Getting a low score from the scale will indicate that their anxiety about the procedure is low.
Fear Means | 1-4 Weeks
  Fear score will be measured with the Children's fear and anxiety scale. The lowest score from the scale can be 0 and the highest score can be 10. As the score obtained from the scale increases, the child's fear increases. In this study, if children score high on the fear section of the scale, it will be determined that their fear of the procedure is high. A low score on the scale will indicate that fears about the procedure are low.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Demir, PhD, Principal Investigator — Hakkari University
Locations (2):
- Turkey (Türkiye) (2):
  - Hakkari University, Hakkâri, Merkez
  - Hakkari University, Hakkâri

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. The data will be shared anonymously if the justification is deemed appropriate.
Supporting Information: Study Protocol
Time Frame: When study will finish, study protocol will share
Access Criteria: It will be shared by the authors.